CLINICAL TRIAL: NCT01472146
Title: Phase II Clinical Trial of Neoadjuvant Treatment With Zolendronic Acid Plus Anthracycline and Taxane in Locally Advanced Breast Cancer
Brief Title: ZoNantax - Zolendronic Acid as Neoadjuvant Therapy Plus Anthracycline and Taxane in Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susanne Crocamo (Other Government)
Responsible Party: Sponsor-Investigator, Susanne Crocamo, Clinical Oncologist, Instituto Nacional de Cancer, Brazil
Organization: Instituto Nacional de Cancer, Brazil (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zo-neo2011
Record Dates: First submitted 2011-09-20; First posted 2011-11-16 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Breast Disease; Neoplasms; Neoplasms by Site
Keywords: Neoadjuvant therapy; Breast cancer HER2 positive; zolendronic acid
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Neoplasms; Neoplasms by Site | interventions — Cyclophosphamide; Docetaxel; Trastuzumab; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zometa neoadjuvant HER2 breast cancer (Experimental): Zo-Nantax arm - Neoadjuvant chemotherapy with association of zoledronic acid and standard treatment with anthracycline followed taxane plus trastuzumab in locally advanced breast cancer HER2 positive HR positive/negative.
  Drug:Cyclophosphamide Drug:Adriamycin Drug:Docetaxel Drug:Trastuzumab Drug:Zolendronic acid
  Interventions: Drug: Zo-Nantax

INTERVENTIONS:
Drug: Zo-Nantax — Experimental:
  AC,Docetaxel,Trastuzumab,Zolendronate
  Drug: AC Adriamycin 60mg/m2 IV plus cyclophosphamide 600mg/m2 every 21 days for 4 cycles
  Drug: Docetaxel
  Docetaxel 100 mg/m2 every 21 days for 4 cycles.
  Drug: Trastuzumab
  Trastuzumab 8mg/kg [loading dose] once then 6mg/kg IV every 21 days for 3 cycles plus docetaxel.
  Drug: zolendronic acid
  Zolendronic acid 4mg IV every 21 days for 8 cycles combine with chemotherapy
  Other Names: Other Names:; Adriblastine RD; Cytoxan; Taxotere®; Herceptin®; Zometa

SUMMARY:
The purpose of this study is to evaluate the association of zoledronic acid with standard treatment with anthracycline followed taxane plus trastuzumab in locally advanced breast cancer HER 2 positive.

DETAILED DESCRIPTION:
This trial combines zolendronic acid with anthracycline followed taxane plus trastuzumab for neoadjuvant treatment of HER 2 positive stage II/III breast cancer.

Zoledronic acid (ZOL) has activity of anti-bone resorption and shows diverse anti-tumor effects in vitro. Some chemical and biological characteristics of ZOL indicate potential for inhibition of tumor growth in pre clinical studies

The primary objective of the study is to evaluate the residual cancer burden (RCB) with the addition of zolendronic acid to standard neoadjuvant therapy. RCB is calculated as a continuous index combining pathologic measurements of primary tumor (size and cellularity) and nodal metastases (number and size). RCB index is a significant predictor of distant relapse-free survival, and can be used to define categories of near-complete response and chemotherapy resistance after neoadjuvant chemotherapy compared with currently used risk factors. Additionally, the study will collect tissue biopsies and blood before and after treatment in order to correlate clinical outcomes with gene expression and radiologic data to predictive response.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIA to IIIB HER-2 positive breast cancer
2. ECOG performance ≤ 2
3. Adequate hematologic function with:

   * Absolute neutrophil count (ANC)> 1500/mm³
   * Platelets ≥ 100.000/mm³
   * hemoglobin ≥ 9g/dL
4. Adequate hepatic and renal function with:

   * Serum bilirubin ≤ 1.5 x the institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤ 2.5 x the institutional upper limit of normal (ULN)
   * Alkaline phosphatase )≤ 2.5 x the institutional upper limit of normal (ULN)
   * Serum creatinine ≤ 1.5 x the institutional upper limit of normal (ULN) or calculated creatinine clearance > 50 mL/min
5. Adequate cardiac function

   * Left ventricular ejection fraction (LVEF)with institutional normal range
6. Knowledge of the investigational nature of the study and ability to provide consent for study participation

Exclusion Criteria:

1. Previous diagnostic of breast or other cancer
2. Pregnancy
3. Metastatic breast cancer
4. Bilateral, synchronous breast cancer
5. Any other disease(s), psychiatric condition, metabolic dysfunction, that contraindicates the use of study drugs or that woud make the patient inappropriate for this study
6. Neuropathy grade > 2 by the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the residual cancer burden (RCB) | 6 months
  Use MD Anderson calculator to quantify the minimal residual disease

SECONDARY OUTCOMES:
Assessing the tolerance to standard neoadjuvant treatment plus zolendronic acid,according to the common toxicity criteria Terminology Criteria for Adverse Events version 3.0. | 6 months
  CTC 4.0
Assessment of the difference in gene expression according to treatment response | 6 months
  Through microarray assays
Prediction of pathological response by MRI calculated from the sequence of apparent diffusion coefficient (ADC) | 4 months
  Make MRI before the start of chemotherapy, after the second cycle and before surgery, and evaluate the changes in the diffusion of water

CONTACTS AND LOCATIONS:
Overall Officials: Susanne C Costa, MD, Principal Investigator — Hospital do Cancer III - INCA
Locations (1):
- Hospital do Cancer III - INCA, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
I don't plan to share IPD